CLINICAL TRIAL: NCT02111213
Title: Virtual Advisors for Physical Activity Promotion in Underserved Communities
Acronym: COMPASS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Northeastern University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Abby C King, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01HL116448 (NIH); R01HL116448 (NIH)
Record Dates: First submitted 2014-04-02; First posted 2014-04-11 (Estimated); Results first posted 2019-10-18 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Sedentary Lifestyle
Keywords: physical activity; Intervention; Attitude to Computers
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The primary study design (involving 245 randomized participants) was a 2-arm non-inferiority randomized trial comparing the effects of physical activity advice delivered by human advisors vs. a computer-based advisor
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Promotora for physical activity (Active Comparator): Weekly sessions with a volunteer promotora at a community center. A promotora is a trained, lay health worker. The promotora will provide guidance, advice and support to participants to encourage them to be more physically active.
  Interventions: Behavioral: Promotora for physical activity
- Carmen system (Experimental): Weekly sessions with the virtual advisor accessed through a computer located at a community center. Carmen is the virtual advisor and will provide guidance, advice and support to participants to encourage them to be more physically active.
  Interventions: Behavioral: Virtual Advisor

INTERVENTIONS:
Behavioral: Virtual Advisor — The virtual advisor is named Carmen. She is an animated, computer-generated figure that speaks to participants and gives advice and support for physical activity.
  Arms: Carmen system
Behavioral: Promotora for physical activity — A promotora is a trained, lay health worker. Promotoras will be trained and supervised to provide advice, support and guidance to people to encourage them to be more physically active. They work with people face to face and by telephone to offer support and advice.
  Arms: Promotora for physical activity

SUMMARY:
The primary aim of this research study is to evaluate the effectiveness of a computer-based 'virtual lay advisor' intervention relative to a proven human lay advisor/promotore intervention to promote regular walking among inactive midlife and older Latino adults. The primary analysis is a non-inferiority analysis comparing these two interventions.

DETAILED DESCRIPTION:
COMPASS (Computerized Physical Activity Support for Seniors) was a single-blind, cluster-randomized noninferiority parallel trial conducted by investigators from Stanford University School of Medicine and Northeastern University. Participants were recruited from community centers in Santa Clara and San Mateo Counties, CA which had been randomized in pairs based on locale to either Virtual or Human advisors. Allocation concealment was accomplished by utilizing staff not directly involved in study enrollment, assessment, or intervention procedures. Both arms received a similar 12-month behavioral PA instruction/support program at their designated community center based on Active Choices-an individually-tailored PA intervention with demonstrated effectiveness and translatability across diverse adult populations. The primary outcome was change in 12-month weekly walking minutes.

In addition to the major trial and primary investigation described above, an exploratory Substudy was conducted separately to begin to evaluate the initial "proof of concept" of a food literacy curriculum in 2 separate community centers that were not part of the major trial. This first-generation exploratory Substudy is not part of the major trial and therefore is not included in this protocol and trial description.

ELIGIBILITY:
Inclusion Criteria:

* Spanish or English-speaking primarily Latino men or women
* Aged greater than or equal to 50 years
* No plans to move within the next year
* Inactive (have not engaged in moderate-intensity or more vigorous physical activity
* > 3 days per week for at least 20 min per day) within last 6 months
* Able to participate in study intervention and assessments at their local neighborhood senior center

Exclusion Criteria:

1. Any medical condition or disorder that would limit participation in moderate intensity physical activity (such as sustained walking), including life-threatening disorders, myocardial ischemia, major functional disabilities in the orthopedic area, or inability to complete baseline assessments for any reason (including psychological, cognitive);
2. Not stable on their medications, including hormone replacement therapy, for ≥ 3 months (given that changes in medications can create additional stress and burden over and above attempts to change lifestyle behaviors);
3. Inability to complete a face-to-face training session with a computer-based program

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abby C King, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Prevention Research Center, Palo Alto, California, United States

REFERENCES:
- [Derived] Zamora AN, Campero MI, Garcia DM, Chavez DM, King AC. Acculturation is associated with 12-month adherence to combined MVPA and sedentary behavior guidelines in a sample of midlife and older Latino/a adults: findings from the COMPASS physical activity trial. BMC Public Health. 2025 Feb 22;25(1):737. doi: 10.1186/s12889-025-21885-3. PMID 39987024
- [Derived] Royer MF, Hauser ME, Zamora AN, Campero MI, Garcia D, Gabaray M, Sheats JL, King AC. Serving up FLAN. a food literacy and nutrition intervention to fend off food insecurity. BMC Nutr. 2024 Jul 23;10(1):102. doi: 10.1186/s40795-024-00909-y. PMID 39044224
- [Derived] Royer MF, Hauser ME, Zamora AN, Campero MI, Garcia D, Gabaray M, Sheats JL, King AC. Serving Up FLAN. A Food Literacy and Nutrition Intervention to Fend Off Food Insecurity. Res Sq [Preprint]. 2024 May 7:rs.3.rs-4331290. doi: 10.21203/rs.3.rs-4331290/v1. PMID 38766254
- [Derived] King AC, Campero MI, Sheats JL, Castro Sweet CM, Hauser ME, Garcia D, Chazaro A, Blanco G, Banda J, Ahn DK, Fernandez J, Bickmore T. Effects of Counseling by Peer Human Advisors vs Computers to Increase Walking in Underserved Populations: The COMPASS Randomized Clinical Trial. JAMA Intern Med. 2020 Nov 1;180(11):1481-1490. doi: 10.1001/jamainternmed.2020.4143. PMID 32986075
- [Derived] King AC, Campero I, Sheats JL, Castro Sweet CM, Garcia D, Chazaro A, Blanco G, Hauser M, Fierros F, Ahn DK, Diaz J, Done M, Fernandez J, Bickmore T. Testing the comparative effects of physical activity advice by humans vs. computers in underserved populations: The COMPASS trial design, methods, and baseline characteristics. Contemp Clin Trials. 2017 Oct;61:115-125. doi: 10.1016/j.cct.2017.07.020. Epub 2017 Jul 22. PMID 28739541
- See also: The Healthy Aging Research and Technology Solutions Lab at Stanford — http://healthyaging.stanford.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Promotora for Physical Activity | Carmen System
Started | 122 | 123
Completed | 116 | 117
Not Completed | 6 | 6
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Promotora for Physical Activity | Carmen System | Total
Number analyzed (Participants) | 122 | 123 | 245
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | NA — Excluded people below 50 years old | NA — Excluded people below 50 years old | NA — Total not calculated because data are not available (NA) in one or more arms.
  Between 18 and 65 years | 92 | 94 | 186
  >=65 years | 30 | 29 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (8.5) | 63.1 (8.3) | 62.8 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 98 | 193
  Male | 27 | 25 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 121 | 120 | 241
  Not Hispanic or Latino | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 122 | 120 | 242
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 122 | 123 | 245
CHAMPS Physical Activity Questionnaire [Mean (Standard Deviation); unit: total weekly walking minutes] | 80.2 (109.3) | 59.6 (84.4) | 70.0 (98.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Weekly Walking Minutes From Baseline to 12 Months
Description: Total weekly walking minutes as measured by self-report (CHAMPS Physical Activity Questionnaire)
Time Frame: baseline, 12 months
Population: 12-month Change in total minutes per week Per protocol
Measure: Mean (Standard Error); unit: minutes per week
Arm/Group | Promotora for Physical Activity | Carmen System
Number analyzed (Participants) | 114 | 117
minutes per week | 134.8 (18.0) | 158.6 (20.1)

2. Secondary Outcome: Change in Sedentary Behavior From Baseline to 12 Months
Description: Self-reported time spent in the following activities: watching television, computer use, reading, socializing, transport and hobbies, and a summary measure (total sedentary time).
Time Frame: baseline, 12 months
Measure: Mean (Standard Error); unit: Minutes per week
Arm/Group | Promotora for Physical Activity | Carmen System
Number analyzed (Participants) | 122 | 123
Minutes per week | -251.9 (110.0) | -272.1 (121.0)

3. Secondary Outcome: Change in Moderate to Vigorous Physical Activity From Baseline to 12 Months
Description: moderate to vigorous intensity physical activity as measured by self-report questionnaire
Time Frame: baseline, 12 months
Measure: Mean (Standard Error); unit: minutes per week
Arm/Group | Promotora for Physical Activity | Carmen System
Number analyzed (Participants) | 122 | 123
minutes per week | 105.4 (13.9) | 103.4 (16.2)

ADVERSE EVENTS:
Time Frame: 1 year for each participant
Arm/Group | Promotora for Physical Activity | Carmen System
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/123
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/123
Other Adverse Events (participants affected / at risk) | 4/122 | 3/123
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Promotora for Physical Activity (N=122) | Carmen System (N=123)
leg pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) — mild leg pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT02111213/Prot_SAP_000.pdf